CLINICAL TRIAL: NCT05425628
Title: European First in Human Study of the NeoChord Transcatheter Mitral Repair System to Assess Safety and Performance in Patients With Symptomatic Mitral Regurgitation
Brief Title: European FIH Study - NeoChord Transcatheter Mitral Repair System for Symptomatic Mitral Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeoChord (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-610710-001
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Prolapse; Degenerative; Mitral Regurgitation; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases
Keywords: NeoChord; Mitral Valve Regurgitation; Mitral Valve Prolapse; Artificial Chordae; Mitral Valve Repair
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, unblinded, single arm first in human/feasibility clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with NeoChord Transcatheter Mitral Repair System (Experimental): Implanting ePTFE sutures as artificial neochordae using NeoChord Transcatheter Mitral Repair System
  Interventions: Device: NeoChord Transcatheter Mitral Repair System (or "NeoChord System")

INTERVENTIONS:
Device: NeoChord Transcatheter Mitral Repair System (or "NeoChord System") — The NeoChord Transcatheter Mitral Repair System is a system of delivery devices and implantable Neochordae and Anchor. The system is designed to percutaneously deliver and deploy the implantable ePTFE sutures, "Neochordae" as artificial chordae at the mitral valve and connect them to the implantable ventricular anchor, "Anchor", using a catheter based system placed into the left side of the heart through the interatrial septum.

SUMMARY:
Safety and performance evaluation of the NeoChord Transcatheter Mitral Repair System in patients with degenerative mitral valve regurgitation.

DETAILED DESCRIPTION:
The objective of this First-in-Human (FIH) evaluation is to assess the safety and performance of the NeoChord Transcatheter Mitral Repair System in treating subjects with symptomatic mitral regurgitation, who are at high risk for standard mitral valve surgery, by using a minimally invasive transcatheter mitral valve repair procedure. The NeoChord Transcatheter Mitral Repair System is indicated for use in patients with grade 3+ or 4+ mitral valve regurgitation who are candidates for surgical mitral valve repair or replacement. The intended purpose for the NeoChord Transcatheter Mitral Repair System is for repair of chordal elongation and rupture resulting in mitral valve prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is 18 to 85 years at time of enrollment.
2. Symptomatic MR (≥3+) confirmed by the echo core lab.
3. Primary segmental prolapse or flail of P2 segment only, or P2 segmental prolapse or flail extending to one adjacent segment (P1 or P3), and the primary regurgitant jet is non- commissural, confirmed by the echo core lab.
4. Leaflet-to-Annulus Index (LAI) ≥ 1.25 based on 2D TEE, confirmed by the echo core lab. (1)
5. Cardiac Index > 2.0.
6. Left Ventricular Ejection Fraction (LVEF) is ≥ 30% (within 90 days prior to subject enrollment based upon TTE).
7. New York Heart Association (NYHA) Functional Class II, III or ambulatory IVa.
8. Subject deemed a high surgical risk per MVARC definition by the site's Heart Team (as a minimum, one cardiac surgeon, one interventional cardiologist, and a cardiac imaging expert).
9. Transseptal catheterization is deemed feasible by the Subject Screening Committee.
10. The subject or the subject's legal representative has been informed of the nature of the study and agrees to its provisions including returning for all follow-up visits and has provided written informed consent.

Exclusion Criteria:

1. MR etiology that is exclusively Secondary (functional).
2. Echocardiographic evidence of EROA ≤ 0.3cm2.
3. Valvular leaflet anatomy or pathology deemed not suitable for the NeoChord Implant.
4. Untreated clinically significant coronary artery disease requiring revascularization.
5. Hypertrophic/restrictive cardiomyopathy, constrictive pericarditis, or other structural heart disease causing heart failure other than cardiomyopathy of either ischemic or non-ischemic etiology.
6. Hypotension (systolic pressure < 90 mmHg)/Cardiogenic shock or other hemodynamic instability requiring theneed for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
7. Fixed pulmonary artery systolic pressure > 2/3 of systemic systolic blood pressure.
8. Evidence of right-sided heart failure with echocardiographic evidence of severe right ventricular dysfunction.
9. Surgical or interventional procedure planned within 30 days prior to index procedure.
10. Prior orthotropic heart transplantation.
11. Life Expectancy < 1 year due to non-cardiac conditions.
12. Chronic Kidney Disease with Creatinine clearance <30 ml/min/1.73m2.
13. Any prior mitral valve surgery or transcatheter mitral valve procedure.
14. Stroke, transient ischemic event, or myocardial infarction within 30 Days prior to index procedure.
15. ModifiedRankinScale>4disability.
16. Class I indication for biventricular pacing (in patient with CRT device not implanted).
17. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator within one month prior to index procedure.
18. Need for cardiovascular surgery (other than MV disease).
19. Aortic or pulmonic valve disease requiring surgery.
20. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
21. Activeendocarditis.
22. Knownseveresymptomaticcarotidstenosis(>70%via ultrasound).
23. Active infections requiring current antibiotic therapy.
24. Active cancer with expected survival < 1 year.
25. Pregnant or planning pregnancy within next 12 months.
26. Currently participating in an investigational drug or another device study.
27. Femoral vein cannot accommodate a 28F catheter or there is evidence of ipsilateral deep vein thrombosis(DVT)).
28. Hepatic insufficiency (MELD > 10).
29. Chronic anemia (Hgb < 9).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The ability of the NeoChord device to be placed without Major Device Related Adverse Events. | 30 days
  * Death (Cardiovascular mortality vs non-cardiovascular);
  * Reintervention (operative or transcatheter) due to progressive or recurrent MR or device related complications;
  * Disabling stroke;
  * Myocardial infarction (MVARC definition);
  * Major access site and vascular complications;
  * Fatal or life-threatening bleeding (MVARC Type III-V);
  * Arrhythmia and conduction disorder requiring permanent pacing;
  * Renal Failure requiring dialysis;
  * Cardiac tamponade.
  All other SAE's and device/procedure-related AE's will be summarized throughout the follow-up duration, as descriptive endpoint data.
NeoChord Technical Success | 30 days
  * Successful access, delivery, and retrieval of the delivery system; and
  * Successful deployment and correct positioning of the implant; and
  * Freedom from emergency surgery or reintervention related to the device or access procedure
  Without any procedural mortality or stroke, at 30-day follow up.

SECONDARY OUTCOMES:
Secondary performance endpoints (MR severity) | 30 days, 90 days, and 180 days post-index procedure
  • Change in LV End diastolic volume index (LVEDVI)
Secondary performance endpoints (MR severity) | 30 days, 90 days, and 180 days post-index procedure
  • Change in LV end-systolic volume index (LVESVI)
Secondary performance endpoints (Patient Success) | 30 days, 90 days, and 180 days post-index procedure
  • Changes in New York Heart Association functional Class (NYHA)
Secondary performance endpoints (Patient Success) | 30 days, 90 days, and 180 days post-index procedure
  • 6-minute walk test distance (6MWT)
Secondary performance endpoints (Patient Success) | 30 days, 90 days, and 180 days post-index procedure
  • Kansas City Cardiomyopathy Questionnaire score (KCCQ)
Secondary performance endpoints (Patient Success) | 30 days
  • Device dysfunction (Central MR grade > 1) follow-up